CLINICAL TRIAL: NCT03021148
Title: Prevalence of Self-reported Gluten Sensitivity in a Population of High-school Students
Brief Title: Self-reported Gluten Sensitivity in High-school Students
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Other Study IDs: ACPM17
Record Dates: First submitted 2016-12-30; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Non-celiac Wheat Sensitivity
Keywords: Non-celiac wheat sensitivity; self-reported
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High-school children: High-school children, age range from 13 to 18 years, from "Liceo Classico" and "Liceo Artistico" "Tommaso Fazello" of Sciacca, Agrigento, Italy
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Administration of questionnaire.

SUMMARY:
It has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have celiac disease or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS). In a previous paper the investigators suggested the term 'Non-Celiac Wheat Sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. To our knowledge, there are very few studies which assessed the prevalence of self-reported gluten-related symptoms in the community and analyze diagnostic outcomes in those referred to secondary gastrointestinal care. In one of these, performed in UK, the authors showed that gluten-related symptoms are self-reported by 13% of the population, with 3.7% consuming a gluten-free diet, despite only 0.8% being aware that they have a formal diagnosis of celiac disease. Of those patients presenting to the gastroenterology department, the majority do not have CD but NCWS. No data are available for boys and girls. Therefore, the aims of this study were 1) to determine the prevalence of self-perceived gluten-sensitivity in a population of high-school students, and 2) to evaluate the demographic and clinical differences between students self-reporting gluten sensitivity and students not reporting food hypersensitivity.

DETAILED DESCRIPTION:
Self-reported food hypersensitivity is common, particularly in women, with a reported prevalence of 20.4% in the UK community. A wide range of gastrointestinal and systemic symptoms may be experienced related to consumption of the intolerant food(s). In addition, patients demonstrate considerably more generalized subjective health complaints in comparison with healthy controls. In this context, it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have celiac disease or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS). In a previous paper the investigators suggested the term 'Non-Celiac Wheat Sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. The clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and extra-intestinal and/or systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). To our knowledge, there are few studies which assessed the prevalence of self-reported gluten-related symptoms in the community and analyze diagnostic outcomes in those referred to secondary gastrointestinal care. In one of these, performed in UK, the authors shown that gluten-related symptoms are self-reported by 13% of the population, with 3.7% consuming a gluten-free diet, despite only 0.8% being aware that they have a formal diagnosis of celiac disease. In this study individuals self-reporting gluten-related symptoms are predominantly female, report an association with IBS, and experience both intestinal and extraintestinal symptoms on gluten ingestion. Of those patients presenting to the gastroenterology department, the majority do not have CD but NCWS. In contrast to the above mentioned data, obtained in adults, no data are available for young people. Therefore, the aims of this study were 1) to determine the prevalence of self-perceived gluten-sensitivity in a population of high-school students, and 2) to evaluate the demographic and clinical differences between students self-reporting gluten sensitivity and students not reporting food hypersensitivity. The students participated in the study by filling out a modified version of a previously validated written questionnaire, to which there were two sections. The first comprised basic demographic information, including age, sex and ethnicity, and a screening section for symptoms consistent with irritable bowel syndrome (IBS) in accordance with the Rome III criteria, also including their past gastrointestinal, psychiatric and allergic history. The second section of the survey enquired for self-reported gluten-related symptoms. Participants were also asked for their use of a gluten-free diet and if they had seen a healthcare professional for their symptoms. A reported diagnosis of celiac disease and wheat allergy in the population group was defined by those who had a doctor diagnosis of celiac disease and wheat allergy and were also taking a gluten-free diet.

ELIGIBILITY:
Inclusion Criteria:

* All students who attended the high-school five-years course, independently by their age.

Exclusion Criteria:

* N/A

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study include high-school children, age range from 13 to 18 years, from "Liceo Classico" and "Liceo Artistico" "Tommaso Fazello" of Sciacca, Agrigento, Italy, evaluated by an ad hoc questionnaire between January 2016 and December 2016.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with self-perceived gluten-sensitivity in a population of high-school students | January 2016 to December 2016
  Number of subjects with self-perceived gluten-sensitivity in a population of high-school students by using an ad hoc questionnaire.

SECONDARY OUTCOMES:
Demographic differences between children self-reporting and children not self reporting gluten-related symptoms | January 2016 to December 2016
  Demographic differences between students self-reporting gluten sensitivity and students not reporting food hypersensitivity
Clinical differences between children self-reporting and children not self reporting gluten-related symptoms | January 2016 to December 2016
  Clinical differences between students self-reporting gluten sensitivity and students not reporting food hypersensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PhD, Study Director — University of Palermo
Locations (2):
- Italy (2):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Department of Internal Medicine, University Hospital of Palermo, Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Carroccio A, D'Alcamo A, Mansueto P. Nonceliac wheat sensitivity in the context of multiple food hypersensitivity: new data from confocal endomicroscopy. Gastroenterology. 2015 Mar;148(3):666-7. doi: 10.1053/j.gastro.2014.11.047. Epub 2015 Jan 24. No abstract available. PMID 25625764
- [Result] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Role of FODMAPs in Patients With Irritable Bowel Syndrome. Nutr Clin Pract. 2015 Oct;30(5):665-82. doi: 10.1177/0884533615569886. Epub 2015 Feb 18. PMID 25694210
- [Result] Young E, Stoneham MD, Petruckevitch A, Barton J, Rona R. A population study of food intolerance. Lancet. 1994 May 7;343(8906):1127-30. doi: 10.1016/s0140-6736(94)90234-8. PMID 7910231
- [Result] Aziz I, Lewis NR, Hadjivassiliou M, Winfield SN, Rugg N, Kelsall A, Newrick L, Sanders DS. A UK study assessing the population prevalence of self-reported gluten sensitivity and referral characteristics to secondary care. Eur J Gastroenterol Hepatol. 2014 Jan;26(1):33-9. doi: 10.1097/01.meg.0000435546.87251.f7. PMID 24216570
- [Result] Sanders DS, Patel D, Stephenson TJ, Ward AM, McCloskey EV, Hadjivassiliou M, Lobo AJ. A primary care cross-sectional study of undiagnosed adult coeliac disease. Eur J Gastroenterol Hepatol. 2003 Apr;15(4):407-13. doi: 10.1097/00042737-200304000-00012. PMID 12655262